CLINICAL TRIAL: NCT06395649
Title: Personalized Pain Treatment by Transcranial Magnetic Stimulation in Patients With Chronic Pain: a Study on Mechanisms
Brief Title: Personalized Treatment by rTMS in Chronic Pain
Acronym: PersoNINpain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Enrico De Martino, Principal investigator, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-20230076
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: When 50% of inclusion is completed, a preplanned interim futility analysis is scheduled to examine safety and the main outcome.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Classical rTMS to M1x (Active Comparator): The patients will receive repetitive transcranial magnetic stimulation (rTMS) to the primary cortex (M1) according to the classical treatment.
  Interventions: Device: Classical rTMS to M1
- High connectivity target (Experimental): The patients will receive repetitive transcranial magnetic stimulation (rTMS) to target showing the largest connectivity during the TMS-EEG assessment one week before starting the treatment
  Interventions: Device: rTMS to the High connectivity target
- Low connectivity target (Experimental): The patients will receive repetitive transcranial magnetic stimulation (rTMS) to target showing the lowest connectivity during the TMS-EEG assessment one week before starting the treatment
  Interventions: Device: rTMS to the low connectivity target
- Sham stimulation (Sham Comparator): Subjects experiencing significant pain reduction (according to the primary outcome) by the treatment will be asked if they would like to continue maintenance stimulation sessions. Participants accepted to join this part of the study will receive 1 stimulation session every 2 weeks for 4 weeks (total of 2 stimulation sessions). The participants will receive either active stimulation exactly as they received previously or sham stimulation with rTMS in a double-blind, randomized, placebo-controlled, two-group setup.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Classical rTMS to M1 — The rTMS intervention consists of 10-Hz rTMS. Thirty trains of ten seconds with an interval of twenty seconds between trains will be delivered, as traditionally performed. Each train includes 100 pulses, and the total number of pulses will be 3,000 given in 15 minutes.
  Arms: Classical rTMS to M1x
Device: rTMS to the High connectivity target — The rTMS intervention consists of 10-Hz rTMS. Thirty trains of ten seconds will be delivered with an interval of twenty seconds between trains. Each train includes 100 pulses, and the total number of pulses will be 3,000 given in 15 minutes. The rTMS will be delivered to the target, showing the highest connectivity.
  Arms: High connectivity target
Device: rTMS to the low connectivity target — The rTMS intervention consists of 10-Hz rTMS. Thirty trains of ten seconds with an interval of twenty seconds between trains will be delivered. Each train includes 100 pulses, and the total number of pulses will be 3,000 given in 15 minutes. The rTMS will be delivered to the target, showing the lowest connectivity.
  Arms: Low connectivity target
Device: Sham rTMS — Sham stimulation was carried out with a sham coil of identical size, color, and shape, emitting a sound similar to that emitted by the active coil.
  Arms: Sham stimulation

SUMMARY:
Previous research has shown the effectiveness of magnetic stimulation of the brain as a supplemental treatment for various conditions, such as depression and chronic pain. However, the application of magnetic stimulation has been standardized across patients without considering individual differences. This one-size-fits-all approach results in only half of the patients benefiting from the treatment, with the other half seeing no improvement in their symptoms. Therefore, a study on individuals with chronic pain will be performed to explore how magnetic stimulation treatments can be tailored to each person. This will involve analyzing brain signal measurements before the start of the therapy and adjusting/personalizing the magnetic stimulations to each individual person.

DETAILED DESCRIPTION:
This project aims to test if the effects of non-pharmacological, non-invasive pain treatment can be enhanced by employing brain connectivity information to guide the application of repetitive transcranial magnetic stimulation (rTMS). Previous efficacy and safety trials have supported that rTMS for pain relief is applied to four main cortical areas: primary motor cortex (M1), dorsolateral prefrontal cortex (DLPFC), anterior cingulate cortex (ACC), and posterosuperior insular (PSI). However, some patients respond to rTMS to one of these targets but not to the others. Since there is no current strategy to know which patient will respond to each treatment target, patients with chronic pain end up undergoing trial and error strategies, which delay their improvement. This is actually not different from challenges related to pharmacological treatment, where each medication only relieves pain in 30-40% of patients, and the choice of each medication is based on "trial-and-error basis".

Several strategies currently aim to provide a more individualized strategy for choosing analgesic interventions based on patient-related information. In order to allow for the design of efficacy trials in the future, the present project is based on a proof-of-concept, mechanistic design. It will employ rTMS stimulation for pain control, but the choice of each of the stimulation targets will be made based on each individual's brain signals as read by EEG recorded before the start of the treatment. Therefore, before receiving a full rTMS treatment, patients will undergo a neurophysiological screening session using single-pulseTMS-EEG. Single-pulseTMS and EEG have been routinely used in the clinic as a part of the neurophysiological assessment of patients for decades but have not yet been used in the association as an attempt to try to guide the choice of treatment. In the screening session, single pulses TMS will be applied to each of the primary network hubs used in therapeutic rTMS: M1, DLPFC, ACC, and PSI. Concomitantly, the EEG oscillatory activity of these four cortical areas will be recorded, and the brain connectivity state will be assessed. By using information derived from a patient´s brain connectivity state using transcranial magnetic stimulation with electroencephalography (TMS-EEG), the most appropriate of the four classic targets will be selected and used in rTMS on an individualized basis. It is hypothesized that the brain regions with low local-to-global connectivity will provide better pain relief compared to non-personalized treatment approaches and compared to targets with optimized local-to-global connectivity status.

A total of 90 subjects with chronic pain will be included in a double-blind, randomized three parallel-arm study comparing the analgesic effect of the therapeutic rTMS target chosen based on TMS-EEG:

1. target area presenting the lowest local-to-global connectivity
2. target area presenting the highest local-to-global connectivity
3. classic M1 stimulation.

The subjects will be allocated in a 1:1:1 ratio to one of three arms (30 subjects per arm). The protocol is designed as an adaptive study, incorporating interim analyses after enrolling 30 and 60 subjects. These evaluations, conducted by a blinded specialist statistician panel, will assess the efficacy of the target selection strategy for each arm, focusing on the primary outcome's progression.

In the initial baseline measurement, the subjects will fill out questionnaires and undergo neurophysiological assessments. After this baseline measurement, the subjects will be assigned to one of the three arms and will receive daily rTMS sessions targeting areas (called induction phase) for 5 consecutive days (Monday to Friday) with either "high connectivity", "low connectivity", or a "classic M1 target". Each of the 5 daily stimulations will last 30 minutes, of which 15 minutes will be under treatment.

The induction phase will be followed by a 6-week maintenance phase, with 1 rTMS session per week (totaling 6 rTMS sessions). At the end of the maintenance phase, primary and secondary outcomes (questionnaires) will be collected to investigate the efficacy of the rTMS treatments. A random subsample of 30 participants (10 from each arm) will be asked if they would like to participate in a second 3-hour neurophysiological assessment to investigate the changes in brain connectivity.

Subjects experiencing significant pain reduction (according to the primary outcome) by the treatment will be asked if they would like to continue maintenance stimulation sessions. Participants accepted to join this part of the study will receive 1 stimulation session every 2 weeks for 4 weeks (total of 2 stimulation sessions). The participants will receive either active stimulation exactly as they received previously or sham stimulation with rTMS in a double-blind, randomized, placebo-controlled, two-group setup. After the extended maintenance phase, primary and secondary outcomes (questionnaires) will be issued, and a random subsample of 20 patients (10 per group) will go through a third, 3-hour-long assessment involving neurophysiological assessment to investigate the changes in connectivity.

When 50% of inclusion is completed, a preplanned interim futility analysis is scheduled to examine safety and the main outcome.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic pain (present most of the days for more than 3 months).
* Pain with a mean pain intensity between 3-9 on a 0-10 pain scale (where 0 means no pain and 10 means the worst pain imaginable).
* Speak and understand English or Danish

Exclusion Criteria:

* Pregnant or breastfeeding
* Current uncontrolled major depression as the main diagnosis
* Current history of substance abuse
* Lack of ability to cooperate, to fully understand the protocol or any difficulty in filling out questionnaires (e.g., due to language or cognitive problems)
* Formal contraindications to TMS application (presence of epilepsy, cranial implanted ferromagnetic devices, e.g., intracranial neurostimulator or cochlear implants, tattoos with metal ink on the face or permanent make up with metal in the face )16
* Unable to answer the "Transcranial Magnetic Stimulation Adult Safety Screen" screening questionnaire.
* Participation in other research protocols within 1 month before the inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (Visual analogue scale) | VAS will be assessed before treatment, after 2 months, and again after 3 months. Responders are those with ≥30% pain reduction at the end of maintenance compared to average pain intensity the week before baseline assessment.
  The '0' represents 'no pain' at all, and '100' represents the 'worst possible pain' that the individual can imagine.

SECONDARY OUTCOMES:
Quality of life (EQ-5D) | Quality of life changes will be investigated before the treatment, immediately after 2 months of treatment, and again after 3 months of treatment.
  EQ-5D is a standardized measure of health-related quality of life
Patients' Global Impression of Change | Patients' Global Impression of Change will be investigated before the treatment, immediately after 2 months of treatment, and again after 3 months of treatment.
  The questionnaire assesses the individual's impression of change after an intervention.
Short Brief Pain Inventory | Short Brief Pain Inventory changes will be investigated before the treatment, immediately after 2 months of treatment, and again after 3 months of treatment.
  9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning.
Short McGill Pain Questionnaire | Short McGill Pain Questionnaire changes will be investigated before the treatment, immediately after 2 months of treatment, and again after 3 months of treatment.
  a comprehensive multidimensional tool that assesses the three main aspects of pain: sensory discriminative, affective-motivational, and cognitive-evaluative
Connectivity analysis | Connectivity changes will be investigated before the treatment, immediately after 2 months of treatment, and again after 3 months of treatment.
  Electroencephalography (EEG) recorded during single pulses of TMS will be used to evaluate brain connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico De Martino, Dr, Principal Investigator — Aalborg University
Locations (1):
- Aalborg University, Gistrup, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No